CLINICAL TRIAL: NCT05618704
Title: A Single Arm, Open Label Intervention Study of a Hydrolyzed Protein Formula to Evaluate Growth, Safety and Tolerance in Infants With a Clinical Diagnosis of Cow's Milk Allergy
Brief Title: Growth, Safety and Tolerance of a Hydrolyzed Protein Infant Formula
Acronym: STORY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SBB21R&38227
Record Dates: First submitted 2022-10-27; First posted 2022-11-16 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Cow Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Intervention Model Description: single arm, open label, interventional, multi-centre study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hydrolyzed protein infant formula (Experimental): All subjects will take the hydrolyzed protein infant formula
  Interventions: Dietary Supplement: Hydrolyzed protein infant formula

INTERVENTIONS:
Dietary Supplement: Hydrolyzed protein infant formula — The subjects will take the formula for 16 weeks

SUMMARY:
This is a single arm, open label, multicenter intervention trial to evaluate growth parameters, cow's milk related symptoms, gastrointestinal tolerance and safety in infants with cow's milk allergy receiving a hydrolyzed protein formula.

DETAILED DESCRIPTION:
The main purpose of this study is to demonstrate adequate growth over a 16-week intervention period in cow's milk allergic infants receiving a hydrolyzed protein formula.

ELIGIBILITY:
Inclusion Criteria:

1. Infants <8 months of age.
2. Infants with a clinical diagnosis of Cow's Milk Allergy (CMA) per local hospital practice, including any of the following criteria:

   1. Based on clinical examination with a careful history, parent-reported symptoms suggestive of CMA, and disappearance of the symptoms when cow's milk was eliminated from the diet for at least two weeks prior to study entry
   2. Based on clinical examination with a careful history, parent-reported symptoms suggestive of CMA, and disappearance of the symptoms while being breastfed with maternal cow's milk protein elimination diet for at least two weeks prior to study entry
   3. History of CoMiSS® score >10 indicating symptoms are likely cow's milk allergic prior to study entry
   4. History of positive result of an oral food challenge with cow's milk prior to study entry
   5. Presence of specific Immunoglobulin E (IgE) to cow's milk protein based on skin prick test (wheel size ≥3mm) or radio-allergosorbent-test (RAST) (>0.7 kilounit per liter (kU/L)) prior to or on the day of study entry.
3. 3. Infants that are still on dairy-derived extensively hydrolysed formula, amino acid-based formula, hydrolysed rice protein formula, soy-based formula or being breastfed by mothers who are on cow's milk protein elimination diet at study entry.
4. Parents / guardians confirm their intention not to administer any products containing cow's milk protein during the study.
5. Expected to consume the specified age-dependent minimum amount of study product per day during the study.
6. Expected to require a milk substitute for CMA management for at least 16 weeks.
7. Written informed consent provided by parents / guardians, according to local law.

Exclusion Criteria:

1. Birth weight-for-age z-score <-2 Standard Deviation (SD) or >+2SD.
2. Infants <37 weeks gestation requiring specific premature formula at the time of study entry.
3. Infants with severe concurrent illness and/or have undergone gastrointestinal surgery such as bowel resection or stoma placement and/or with Down syndrome or other syndromes where functional gastrointestinal disorders are common.
4. Infants that are more suitable to use Amino Acid Formula (AAF) as first-line formula, including but not limited to those with high risk of anaphylaxis (prior history of anaphylaxis and currently not using extensively Hydrolysed Formula (eHF)), faltering growth / failure to thrive, or severe forms of non-IgE-mediated CMA such as eosinophilic oesophagitis, enteropathies, or Food Protein-Induced Enterocolitis Syndrome (FPIES).
5. Infants with diagnosis of rice allergy or known allergy to any of the ingredients in the study product.
6. Investigator's uncertainty about the willingness or ability of the parents / guardians to comply with the protocol requirements.
7. Participation in any other studies involving investigational or marketed products concomitantly or within two weeks prior to entry into the study.

Ages: 0 Days to 8 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2023-03-16 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
Adequate growth | 16 weeks
  Proportion of subjects with growth classified as adequate (by interpreting WHO z-scores weight-for-age and weight-for-length)

OTHER OUTCOMES:
Growth | 16 weeks
  Weight, length, head circumference, BMI and corresponding World health Organization (WHO) z-scores
Cow's milk related symptoms | 16 weeks
  CoMiSS and parent completed diary
Gastrointestinal tolerance | 16 weeks
  Parent completed diary, incidence of gastrointestinal adverse effects. Tolerance will be evaluated on the basis of the number of gastrointestinal events including diarrhea, constipation, bloating, distension, nausea, vomiting, burping, flatulence and regurgitation and abdominal discomfort or pain reported for subjects during their participation in the study.
Concentration of markers of mineral status in blood | 16 weeks
  * Zinc (Zn)
  * Calcium (Ca)
  * Phosphate (P)
  * Ferritin (Fe)
  * Magnesium (Mg)
Study product intake (ml/day) and complementary foods/drinks (food diary) | 3 days prior to the last visit
  Parent completed diary
Study product appreciation | 16 weeks
  Parent completed questionnaire (questions with scales e.g., strongly agree - strongly disagree)

CONTACTS AND LOCATIONS:
Locations (1):
- Promed Medical Centre, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No